CLINICAL TRIAL: NCT00851188
Title: Internet Delivered Self-help for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaap Lancee (Other)
Responsible Party: Sponsor-Investigator, Jaap Lancee, PhD, Utrecht University
Organization: Utrecht University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UU-vandenBout
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- internet CBT self-help (Experimental): CBT via the internet
  Interventions: Behavioral: Internet CBT self-help
- CBT self-help booklet (Experimental)
  Interventions: Behavioral: CBT self-help booklet
- Waiting list (Active Comparator)
  Interventions: Other: Waiting list

INTERVENTIONS:
Behavioral: Internet CBT self-help — Internet based Cognitive behavioral self-help method for insomnia
  Arms: internet CBT self-help
Behavioral: CBT self-help booklet — Cognitive behavioral self-help method for insomnia via booklet
  Arms: CBT self-help booklet
Other: Waiting list — Waiting list
  Arms: Waiting list

SUMMARY:
The current study aims to evaluate the effects of internet-delivered self-help CBT for insomnia through a randomised controlled trial. Adult persons with insomnia will be invited via a popular scientific website to fill out online questionnaires. Participants will be randomised into treatment groups or the waiting list. Participants will be measured 4, 16, and 40 weeks after intervention with the same questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia
* Access to the internet

Exclusion Criteria:

* Alcohol or substance abuse
* Severe depression
* Being suicidal
* Sleep apnea
* Schizophrenic or having a psychosis disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Sleep Diary | 1 year
  Daily self-observation used to calculate Total Sleep Time, Wake After Sleep Onset, Sleep Onset Latency, Sleep Efficiency, and Day ratings.

SECONDARY OUTCOMES:
Anxiety rating | 1 year
  Measured with the HADS
Depression ratings | 1 year
  Measured with the CES-D
Sleep medication | 1 year
  Measured in the daily diary log

CONTACTS AND LOCATIONS:
Locations (1):
- Utrecht University, Utrecht, Utrecht, Netherlands

REFERENCES:
- See also: Popular-Scientific website about insomnia — http://www.insomnie.nl